CLINICAL TRIAL: NCT05797831
Title: A Phase 2/3 Study of Navtemadlin as Maintenance Therapy in Subjects With TP53WT Advanced or Recurrent Endometrial Cancer Who Responded to Chemotherapy
Brief Title: Study of Navtemadlin as Maintenance Therapy in TP53WT Advanced or Recurrent Endometrial Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kartos Therapeutics, Inc. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRT-232-118; ENGOT en-21 (Other: ENGOT); GOG-3089 (Other: GOG Foundation)
Record Dates: First submitted 2023-03-07; First posted 2023-04-04 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Cancer
Keywords: navtemadlin
MeSH Terms: conditions — Endometrial Neoplasms | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Arm 1 (Experimental): Navtemadlin administered orally at 180 mg, once daily (QD) on Days 1-7 in a 28-day treatment cycles.
  Interventions: Drug: Navtemadlin
- Part 1 Arm 2 (Experimental): Navtemadlin administered orally at 240 mg, once daily (QD) on Days 1-7 in a 28-day treatment cycles.
  Interventions: Drug: Navtemadlin
- Part 1 Arm 3 (No Intervention): Observational control ("watch and wait") on a 28-day cycle.
- Part 2 Arm A (Experimental): Navtemadlin administered orally at 180 mg once daily (QD) on Days 1-7 in a 28-day treatment cycles.
  Interventions: Drug: Navtemadlin
- Part 2 Arm B (Experimental): Navtemadlin administered orally at 240 mg once daily (QD) on Days 1-7 in a 28-day treatment cycles.
  Interventions: Drug: Navtemadlin
- Part 2 Arm C (Placebo Comparator): Placebo administered orally at 180 mg once daily (QD) on Days 1-7 in a 28-day administration cycle.
  Interventions: Drug: Navtemadlin Placebo
- Part 2 Arm D (Placebo Comparator): Placebo administered orally at 240 mg once daily (QD) on Days 1-7 in a 28-day administration cycle.
  Interventions: Drug: Navtemadlin Placebo

INTERVENTIONS:
Drug: Navtemadlin — Navtemadlin is an experimental MDM2 anticancer drug taken by mouth
  Other Names: KRT-232
  Arms: Part 1 Arm 1; Part 1 Arm 2; Part 2 Arm A; Part 2 Arm B
Drug: Navtemadlin Placebo — Navtemadlin placebo is a placebo that is the same in appearance to navtemadlin drug taken by mouth
  Arms: Part 2 Arm C; Part 2 Arm D

SUMMARY:
This study evaluates navtemadlin as maintenance treatment for patients with advanced or recurrent endometrial cancer (EC) who have achieved complete response or partial response on chemotherapy.

The study will be conducted in 2 parts. Part 1 will evaluate safety and efficacy of two different doses of navtemadlin alongside an observational control arm to determine the Phase 3 navtemadlin dose. Part 2 will evaluate the efficacy and safety of navtemadlin Phase 3 dose compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1
* Histologically or cytologically confirmed diagnosis of endometrial cancer documented as TP53WT
* Subjects with advanced or recurrent disease must have completed a single line of up to 6 cycles of taxane-platinum based chemo and achieved a CR or PR per RECIST V1.1
* Adequate hematologic, hepatic and renal function (within 14 days)

Exclusion Criteria:

* Has any sarcomas or small-cell carcinomas with neuroendocrine differentiation
* Prior immune therapy, cytokine therapy, or any investigational therapy (within 28 days)
* Indwelling surgical drains
* Grade 2 or higher QTc prolongation
* History of major organ transplant
* History of bleeding diathesis; major hemorrhage or intracranial hemorrhage (within 24 weeks)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: To determine the navtemadlin Phase 3 dose | 12 months
  Safety review committee (SRC) will determine the navtemadlin Phase 3 dose for Part 2 based on safety data from Part 1
Part 2: To compare progression-free (PFS) survival by independent review committee (IRC) between navtemadlin and placebo | 50 months
  PFS defined as the time from randomization to disease progression by IRC or death, whichever occurs first

SECONDARY OUTCOMES:
Part 1: To evaluate the treatment effect of navtemadlin on PFS by IRC and investigator assessment | 50 months
  PFS defined as the time from randomization to disease progression by IRC/investigator assessment or death, whichever occurs first
Part 2: To evaluate the treatment effect of navtemadlin on the time to first subsequent treatment (TFST) | 50 months
  TFST defined as the time from randomization to initiation of first subsequent anticancer therapy or death, whichever occurs first
Parts 1 and 2: To determine the pharmacokinetic (PK) profile of navtemadlin | 1 day
  Will determine the Maximum observed concentration (Cmax)
Parts 1 and 2: To determine the pharmacokinetic (PK) profile of navtemadlin | 1 day
  Will determine the area under the plasma concentration versus time curve (AUC)
Parts 1 and 2: To determine the pharmacokinetic (PK) profile of navtemadlin | 1 day
  Will determine the time of maximum plasma concentration (Tmax)
Parts 1 and 2: To evaluate the treatment effect of navtemadlin on the disease control rate (DCR) | 50 months
  Best response of complete response (CR), partial response (PR) or stable disease (SD) by IRC/investigator assessment among subjects with PR as best response from prior chemotherapy

CONTACTS AND LOCATIONS:
Locations (83):
- United States (19):
  - Kaiser Permanente Center, Vallejo, California
  - Northside Hospital, Atlanta, Georgia
  - St. Joseph, Savannah, Georgia
  - Dr. Sudarshan K. Sharma, Ltd., Hinsdale, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - FirstHealth Carolinas, Pinehurst, North Carolina
  - OhioHealth Institute, Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-San Antonio Medical Center, San Antonio, Texas
- Austria (3):
  - University Hospital Graz, Department of Gynecology and Obstetrics, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Canada (2):
  - Cross Cancer Institute, Edmonton
  - CHUM - University of Montreal Hospital Centre, Montreal
- Odense University Hospital, Odense, Denmark
- Tartu University Hospital, Tartu, Estonia
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Turku University Hospital, Turku
- Georgia (3):
  - LTD High Technology hospital Medcenter, Batumi
  - American Hospital Network LLC, Tbilisi
  - Caucasus Medical Centre, Tbilisi
- Hungary (2):
  - National Institute of Oncology, Budapest
  - University of Debrecen Clinical Center, Debrecen
- Israel (3):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (13):
  - A.O. Cannizzaro, Catania
  - IRCCS Istituto Romangolo per lo Studio dei Tumori "Dino Amadori", Forlì
  - Ospedale Policlinico San Martino, Genoa
  - ASST di Lecco-Ospedale Alessandro Manzoni, Lecco
  - Ospedale San Luca, Lucca
  - Osp. Niguarda, Milan
  - University Hospital of Parma, Parma
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Ospedale di Prato S. Stefano, Prato
  - Ospedale Santa Maria delle Croci, Ravenna
  - "Azienda Unità Sanitaria Locale della Romagna - Hospital ""Infermi"" of Rimini Oncology Department", Rimini
  - Policlinico Umberto, Rome
  - Ospedale Filippo Del Ponte, Varese
- Lithuania (2):
  - Health Sciences Kaunas Clinics, Kaunas
  - Nation Cancer Institute of Lithuania, Vilnius, Vilnius
- Norway (3):
  - Southern Hospital Sorlandet, Kristiansand
  - Oslo University Hospital HF, Oslo
  - Sykehusapotek Nord Tromsø, Tromsø
- Poland (9):
  - Białostockie Centrum Onkologii, Bialystok
  - Szpitale Pomorskie, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NIO-PIB Oddzial w Gliwicach, Gliwice
  - Centrum Badań klinicznych Jagiellońskie Centrum Innowacji, Krakow
  - Siedleckie Centrum Onkologii, Olsztyn
  - Uniwersytecki Szpital, Poznan
  - NIO-PIB Klinika Gine-Onk, Warsaw
  - Lower Silesian Oncology, Pulmonology and Hematology Center, Department of Oncological Gynecology, Wroclaw
- Romania (7):
  - Bucharest CF2 Hospital, Bucharest
  - Ovidius Clinical Hospital SRL, Constanța
  - Onco Clinic Consult S.A., Craiova
  - Oncology Center "Sf. Nectarie", Craiova
  - Gral Medical S.R.L. - Oncofort Hospital, Piteşti
  - Oncocenter, Oncology Clinic SRL, Timișoara
  - SC Oncomed SRL, Timișoara
- Slovenia (2):
  - Institute of Oncology Ljubljana, Ljubljana
  - University Clinical Center Maribor, Maribor
- Spain (9):
  - CHUAC (Hospital de Coruña), A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Galdakao-Usansolo, Galdakao
  - Hospital Universitario de Jaen, Jaén
  - H.G.U. Jerez de la Frontera, Jerez de la Frontera
  - Hospital U Insular de GC, Las Palmas
  - Hospital de Leon, León
  - HCU Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario de Valme, Seville
- Sweden (2):
  - Linkoping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm